CLINICAL TRIAL: NCT07075042
Title: Comparing the Attentional Demands and Functional Outcomes of Pattern Recognition and Direct Myoelectric Control in People With Transradial Amputation
Brief Title: Comparing the Attentional Demands and Functional Outcomes in People With Transradial Amputation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM20029330
Record Dates: First submitted 2025-06-11; First posted 2025-07-20 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Amputation
Keywords: Transradial Amputation; Direct Myoelectric Control; Pattern Recognition

STUDY DESIGN:
Intervention Model Description: 6-month crossover trial with current upper limb prosthesis users. The intervention condition in this study is PRC arm controller method. The control condition is DC, the standard-of-care, two-site controller strategy used in most myoelectric prostheses. Participants in the study will be provided with a transradial prosthesis featuring a wrist unit and a multi-function hand as part of this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRC arm controller method intervention first and then the DC intervention (Active Comparator): This arm will have the PRC arm controller method intervention first. The intervention condition in this study is PRC arm controller method. The control condition is DC, the standard-of-care, two-site controller strategy used in most myoelectric prostheses. Participants in the study will be provided a transradial prosthesis with a wrist unit and multi-function hand as part of this study.
  Interventions: Device: Training with PRC; Device: Training with DC; Device: PRC Device use in community and home; Device: DC Device use in community and home
- the DC intervention first and then the PRC arm controller method intervention (Active Comparator): This arm will have the DC arm (standard of care) intervention first.The intervention condition in this study is PRC arm controller method. The control condition is DC, the standard-of-care, two-site controller strategy used in most myoelectric prostheses. Participants in the study will be provided a transradial prosthesis with a wrist unit and multi-function hand as part of this study.
  Interventions: Device: Training with PRC; Device: Training with DC; Device: PRC Device use in community and home; Device: DC Device use in community and home

INTERVENTIONS:
Device: Training with PRC — All participants will receive in-person training with an onsite study prosthetist for the assigned controller strategy. The purpose of the training will be to instruct users on the care of the device formally and to achieve a basic level of functional performance. Training will be individualized according to clinical discretion consistent with clinical practice. Training will consist of up to four sessions to facilitate participants' use of the assigned controller system. The number of sessions will be competency-based (i.e., determined by the ability of each participant to explain or perform specified tasks). A standardized protocol and training checklist have been developed by clinical subject matter experts (i.e., upper limb prosthetists and occupational therapists).
Device: Training with DC — All participants will receive in-person training with an onsite study prosthetist for the assigned controller strategy. The purpose of the training will be to instruct users on the care of the device formally and to achieve a basic level of functional performance. Training will be individualized according to clinical discretion consistent with clinical practice. Training will consist of up to four sessions to facilitate participants' use of the assigned controller system. The number of sessions will be competency-based (i.e., determined by the ability of each participant to explain or perform specified tasks). A standardized protocol and training checklist have been developed by clinical subject matter experts (i.e., upper limb prosthetists and occupational therapists).
Device: PRC Device use in community and home — After the training sessions, all subjects will use the PRC device in their homes, just in a different order.
Device: DC Device use in community and home — After the training sessions, all subjects will use the DC device in their homes, just in a different order

SUMMARY:
Regular prosthesis use by an individual with upper limb loss can help improve general well-being. Individuals who do not use their prosthesis report more significant functional disability and lower health-related quality of life. A significant proportion of individuals with upper limb loss report high levels of disuse or discontinued use of their prosthesis because of physical pain or psychological distress, perceptions that the device provides no functional benefit, undesirable aesthetics, and issues with fit, comfort, weight, or design of their prosthetic device. Being able to exert intuitive control over a device would theoretically pose a lower cognitive burden to the user, concomitantly increasing functional performance. This effect could bolster device use and satisfaction.

DETAILED DESCRIPTION:
Pattern recognition controller (PRC) systems for upper limb prostheses are a replacement to conventional direct controller (DC) systems. For decades, two-site DC has been the primary method for controlling upper limb myoelectric prosthetic devices. The DC method involves recording surface electromyography (EMG) at two 'control sites', ideally an antagonistic muscle pair in the residual limb. Alternatively, PRC is an emerging approach to myoelectric control that can potentially address the key limitations of DC. PRC uses pattern classifiers to discern intended motions based on EMG signals recorded from multiple sites on the residual limb. PRC combines EMG signals captured from multiple electromyography sensors on the residual limb to determine control intent and subsequently translate that intent to the wrist and hand/terminal device unit, while DC relies on signal level from two sensors, with the dominant signal being translated into a movement intention to control the prosthesis. The PRC technique avoids the need to isolate muscle activations and non-intuitive triggers. PRC offers a potentially more natural and intuitive way to operate along a greater range of motion, as well as perform a larger number of hand grasps when compared to DC - particularly during tasks that are complex and require rapid switching between actions of the wrist and/or terminal device. PRC also allows the user to recalibrate control at any time, better accommodating day-to-day variations in socket fit and positioning of the electrodes over the targeted muscle sites. While both systems have been commercially available for more than a decade or more, there is lack of comparative evidence to inform clinical decisions and guide policy. The current trial will investigate potential functional advantages and disadvantages of PRC compared to DC.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Unilateral transradial limb loss
* At least 6 months since loss
* Previous or current use of a myoelectric device for 3 months or longer
* Use of a prosthesis at least 4 days each week
* Ability to read, write, and understand English
* Willingness to use each control strategy as primary device for 3 months each (6 months commitment total)

Exclusion Criteria:

* Any health condition that would prevent safely completing trial activities
* Discontinued use of a myoelectric prosthesis due to non-financial reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Clothespin Relocation Test (CRT) | 6 months (During the course of the study procedures/participation)
  The CRT measures upper limb prosthesis performance. The test requires participants to rotate each clothespin 90° before placing it onto the vertical bar, which necessitates use of more than one joint motion. Faster completion times are indicative of superior prosthesis control and dexterity. This will be completed under single-task and dual-task conditions.

SECONDARY OUTCOMES:
Brief Activity Measure for Upper Limb Amputees (BAM-ULA) | 6 months (During the course of the study procedures/participation)
  The BAM-ULA measures an upper limb prosthesis user's ability to perform daily functional activities, including both unimanual and bimanual tasks. This outcome measure requires the participant to tuck their shirt into the back of their pants, place a 20-pound bag on a shelf, open a sealed water bottle and drink from it, remove a wallet from their back pocket, put wallet into their back pocket, take a gallon jug out of the refrigerator, open and pour with the jug, brush their hair, use a fork, and open a door with a doorknob. This outcome measure is scored based on task completion. A higher composite score is indicative of superior prosthesis control.
Jebsen-Taylor Hand Function Test (JTHF) | 6 months (During the course of the study procedures/participation)
  The JTHF is a standardized measure that tests an individual's unimanual hand function for completing activities of daily living. This test requires the participant to write, turn cards over, pick up and manipulate small objects, simulate feeding, stack checkers, and pick up lighter and heavier larger objects. Faster completion times are indicative of superior prosthesis control and hand function.
Orthotic and Prosthetic Users Survey (UEFS-P) | 6 months (During the course of the study procedures/participation)
  The UEFS-P measures functional status, quality of life, and satisfaction with devices and services among those receiving orthotic and prosthetic care. Participants will respond to 29 items. Higher scores reflect greater perceived function.
Patient Experience Measure (PEM) | 6 months (During the course of the study procedures/participation)
  The PEM measures social interaction, self-efficacy, embodiment, intuitiveness, wellbeing, and self-consciousness of upper limb prosthesis users. Higher scores reflect increased ability.
Prosthesis Task Load Index (PROS-TLX) | 6 months (During the course of the study procedures/participation)
  The PROS-TLX assesses the mental, physical, and emotional demands of using a prosthesis. The PROS-TLX is designed to rate the demand after a specified task is immediately finished. Participants will complete the measure after finishing the performance tests. Higher ratings are indicative of lower mental, physical, or emotional demands.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Darter, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States